CLINICAL TRIAL: NCT01389700
Title: A Randomized, Double-blind, Placebo-controlled Trial to Assess the Pharmacokinetics, Pharmacodynamics and Safety of a Single Dose of SAR279356 in Patients Hospitalized in Intensive Care Unit and on Mechanical Ventilation
Brief Title: Pharmacokinetics, Pharmacodynamics and Safety Evaluation of SAR279356 in Intensive Care Unit Mechanically Ventilated Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in patient recruitment in the participating sites
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PKD11791; U1111-1118-6717 (Other: UTN)
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-11

CONDITIONS: Infection Prophylaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- SAR279356 dose 1 (Experimental): SAR279356 dose 1, single administration
  Interventions: Drug: SAR279356
- SAR279356 dose 2 (Experimental): SAR279356 dose 2, single administration
  Interventions: Drug: SAR279356
- Placebo (Placebo Comparator): Matching placebo, single administration
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SAR279356 — Pharmaceutical form: solution for infusion
  Route of administration: intravenous infusion
  Arms: SAR279356 dose 1; SAR279356 dose 2
Drug: placebo — Pharmaceutical form: solution for infusion
  Route of administration: intravenous infusion
  Arms: Placebo

SUMMARY:
Primary Objective:

- To determine the pharmacokinetics (PK) of a single intravenous (IV) dose of SAR279356 administered to intensive care unit (ICU) patients on mechanical ventilation

Secondary Objectives:

* To determine the safety and tolerability of SAR279356
* To evaluate the pharmacodynamics (PD) and immunogenicity of SAR279356
* Exploratory efficacy of SAR279356 on prevention of bacterial infections

DETAILED DESCRIPTION:
Total study duration (from screening to last follow-up visit) is 91 days break down as follows:

* Screening: 1 day prior to dosing;
* Treatment period: one IV injection on Day 1;
* Follow-up period: 90 days

ELIGIBILITY:
Inclusion criteria :

* ICU patients on mechanical ventilation at the time of randomization
* Patients or legally authorized representative (LAR) giving written informed consent.

Exclusion criteria:

* Patients <18 years of age;
* Documented Pseudomonas infection or colonization in the last 30 days;
* Immunocompromised patients
* Hypersensitivity to the study drug and/or to prior therapy with monoclonal antibodies;
* Patient who has taken other investigational drugs or prohibited therapy for this study within 1 month or 5 half-lives, whichever is longer;
* Patient or LAR who withdraws consent during the screening (starting from signed informed consent form);
* Acute liver injury related criteria at the time of study entry:
* Pregnant or breast-feeding women

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters of SAR279356 : Ceoi, AUClast and CL | 90 days

SECONDARY OUTCOMES:
Opsonophagocytic assay (OPA) | 90 days
Opsonophagocytic killing assay (OPK) | 90 days
Dosage of human anti-human antibodies (HAHA) | 90 days
Occurrence of infections | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- United States (6):
  - Investigational Site Number 840010, Los Angeles, California
  - Investigational Site Number 840020, Stanford, California
  - Investigational Site Number 840006, Jacksonville, Florida
  - Investigational Site Number 840001, Pikeville, Kentucky
  - Investigational Site Number 840009, Butte, Montana
  - Investigational Site Number 840003, Camden, New Jersey